CLINICAL TRIAL: NCT00003039
Title: A Phase II Trial of Flavopiridol (NSC 649890) Administered as a 72-Hour Continuous Infusion Every 2 Weeks in Patients With Previously Treated Intermediate and High Grade Non-Hodgkin's Lymphoma Including Mantle Cell Lymphoma
Brief Title: Flavopiridol in Treating Patients With Recurrent Intermediate-Grade or High-Grade Non-Hodgkin's Lymphoma or Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02253; UCCRC-8548; NCI-T96-0099; CDR0000065663 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2000-04

CONDITIONS: Lymphoma
Keywords: recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell | interventions — alvocidib

ARMS (1):
- Arm I (Experimental): Patients receive treatment on an outpatient basis. Flavopiridol is administered as a continuous infusion over 72 hours every 2 weeks. Patients receive a minimum of 4 cycles of therapy unless unacceptable toxicity or disease progression occurs.
  Interventions: Drug: alvocidib

INTERVENTIONS:
Drug: alvocidib

SUMMARY:
Phase II trial to study the effectiveness of flavopiridol in treating patients with recurrent intermediate-grade or high-grade non-Hodgkin's lymphoma or mantle cell lymphoma. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective response rate to flavopiridol by patients with previously treated intermediate and high grade non-Hodgkin's lymphoma and mantle cell lymphoma.

II. Determine the toxicity of flavopiridol administered as a continuous infusion every 2 weeks in these patients.

III. Study the pharmacokinetics of flavopiridol in these patients.

OUTLINE: This is an open label, multi-institutional study.

Patients receive treatment on an outpatient basis. Flavopiridol is administered as a continuous infusion over 72 hours every 2 weeks. Patients receive a minimum of 4 cycles of therapy unless unacceptable toxicity or disease progression occurs. Patients are followed until death.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intermediate or high grade non-Hodgkin's lymphoma (NHL) and mantle cell lymphoma with clinical or pathological evidence of recurrent disease
* Measurable or evaluable disease
* CNS metastases not requiring intravenous steroid therapy allowed

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: CALGB 0-2
* Life expectancy: At least 12 weeks
* Absolute neutrophil count at least 1500/mm3 (unless due to bone marrow involvement by lymphoma)
* Platelet count at least 100,000/mm3 (unless due to bone marrow involvement by lymphoma)
* At least 7 days since platelet transfusion
* Hemoglobin at least 9.0 g/dL
* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL OR creatinine clearance at least 60 mL/min
* No significant uncontrolled medical or psychiatric illness
* No active serious infection
* Not pregnant or lactating
* Fertile patients must use effective contraception
* Central venous catheter required prior to study entry

PRIOR CONCURRENT THERAPY:

* No more than 1 prior chemotherapy regimen
* At least 4 weeks since prior chemotherapy and recovered from all toxic effects Prior chemotherapy must contain anthracycline if intermediate or high-grade NHL other than mantle cell
* No concurrent treatment with other chemotherapeutic or investigational antineoplastic drugs
* At least 4 weeks since prior radiation therapy and recovered (Site of only measurable disease must not be located within prior radiation therapy port)
* No concurrent radiation therapy to any lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1997-09; Primary Completion 2000-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Zimmerman, MD, Study Chair — University of Chicago
Locations (10):
- United States (10):
  - Clinical Sciences Building, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana